CLINICAL TRIAL: NCT00986037
Title: Assessment of the Safety of ABT-308 in Healthy Volunteers and Subjects With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Catherine Tripp MD PhD, Abbott
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: M10-378
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2011-03

CONDITIONS: Asthma
Keywords: Adverse events; Pharmacokinetics
MeSH Terms: conditions — Asthma | interventions — cendakimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- IV ABT-308 in asthmatics (Experimental): ABT-308 single escalating doses in mild to moderate asthmatics
  Interventions: Drug: ABT-308; Drug: Placebo
- SC ABT-308 in asthmatics (Experimental): ABT-308 multiple SQ doses in mild to moderate asthmatics
  Interventions: Drug: ABT-308; Drug: Placebo
- IV ABT-308 in healthy volunteers (Experimental): ABT-308 single escalating IV doses in healthy volunteers
  Interventions: Drug: ABT-308; Drug: Placebo

INTERVENTIONS:
Drug: ABT-308 — Single IV doses
  Arms: IV ABT-308 in asthmatics; IV ABT-308 in healthy volunteers
Drug: ABT-308 — Multiple SC doses x 3
  Arms: SC ABT-308 in asthmatics
Drug: Placebo — Single IV dose
  Arms: IV ABT-308 in asthmatics; IV ABT-308 in healthy volunteers
Drug: Placebo — Multiple SC doses x 3
  Arms: SC ABT-308 in asthmatics

SUMMARY:
The primary purpose of this study is to determine the safety, tolerability and pharmacokinetics of ABT-308 in healthy volunteers and patients with mild to moderate controlled asthma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:

  1. A condition of good health based upon the results of medical history, physical examination, vital signs, laboratory profile and ECG.
  2. BMI 18 to 29, inclusive.
* Mild asthma patients:

  1. Diagnosis of well-controlled, mild to moderate asthma by GINA guidelines for > or = to 6 months
  2. A condition of good health (than mild to moderate asthma) based upon the results of medical history, physical examination, vital signs laboratory profile and EDG.
  3. BMI 18 to 34, inclusive.

Exclusion Criteria:

1. Asthma exacerbation within 8 weeks of Study Day 1.
2. Clinically significant allergic reaction to any drug, biologic, food, or vaccine.
3. History of allergic reaction or significant sensitivity to constituents of study drug.
4. Receipt of any investigational product within 30 days or 5 half-lives (whichever is longer) prior to study drug administration.
5. Subject is a smoker or has a history of smoking within the 6-month period preceding study drug administration.
6. Current enrollment in another clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be determined by evaluation of adverse events, vital sign monitoring, physical examination, electrocardiograms, lung function and laboratory assessments. | 12 weeks after last dose

SECONDARY OUTCOMES:
Pharmacokinetics will be determined by measuring serum concentration of ABT-308. | 12 weeks after last dose
Immunogenicity will be determined by measuring serum concentrations of anti-ABT-308 antibodies. | 12 weeks after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Campbell, MD, Study Director — Abbott

REFERENCES:
- [Result] Tripp CS, Cuff C, Campbell AL, Hendrickson BA, Voss J, Melim T, Wu C, Cherniack AD, Kim K. RPC4046, A Novel Anti-interleukin-13 Antibody, Blocks IL-13 Binding to IL-13 alpha1 and alpha2 Receptors: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation First-in-Human Study. Adv Ther. 2017 Jun;34(6):1364-1381. doi: 10.1007/s12325-017-0525-8. Epub 2017 Apr 28. PMID 28455782